CLINICAL TRIAL: NCT05404360
Title: A Prospective Double Blind Randomized Controlled Trial to Evaluate the Long Term Efficacy and Durability of the BrainsWay Deep Transcranial Magnetic Stimulation (Deep TMS) in Obsessive-Compulsive Subjects
Brief Title: Evaluation of the Long Term Efficacy and Durability of the BrainsWay Deep TMS in OCD Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTP-OCD-02
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: The BrainsWay Deep TMS device is intended to be used as an adjunct for the treatment of adult patients suffering from Obsessive-Compulsive Disorder (OCD). The device technology is based on the application of deep brain TMS by means of repetitive pulse trains at a predetermined frequency.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The treatment administrator, all study personnel and patients will be blinded to the treatment being administrated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Group (Experimental): During the acute treatment phase, subjects will receive daily prefrontal Deep TMS treatment, 5 days a week for 6 consecutive weeks. Following the acute phase, patients will receive semi-weekly Deep TMS stimulation for an additional seven weeks. Treatment will include a total of 44 treatments over 13 weeks.
  Interventions: Device: BrainsWay Deep TMS HAC/H7-Coil
- Sham Control Group (Sham Comparator): During the acute treatment phase, subjects will receive daily prefrontal sham treatment, 5 days a week for 6 consecutive weeks. Following the acute phase, patients will receive semi-weekly sham stimulation for an additional seven weeks. Treatment will include a total of 44 treatments over 13 weeks.
  Interventions: Device: BrainsWay Deep TMS Sham Coil

INTERVENTIONS:
Device: BrainsWay Deep TMS HAC/H7-Coil — The BrainsWay HAC/H7-Coil Deep TMS System is composed of four main components: an electromagnetic H7/HAC-Coil, TMS stimulator, cooling system and positioning arm.
  Other Names: Active Treatment
  Arms: Treatment Group
Device: BrainsWay Deep TMS Sham Coil — The experimental system has two coils in the same helmet, a sham and active coil.
  The sham coil has a similar acoustic artifact as the active coil and it administers a superficial stimulation to maintain blinding. The system assigns the active or sham coil based on the patient ID during the high frequency treatment.
  Arms: Sham Control Group

SUMMARY:
A Prospective Double Blind Randomized Controlled Trial to Evaluate the Long Term Efficacy and Durability of the BrainsWay Deep Transcranial Magnetic Stimulation (Deep TMS) in Obsessive-Compulsive Subjects

DETAILED DESCRIPTION:
The study is a randomized, double-blind, multi-center trial comparing active Deep TMS treatment to sham treatment over the course of the trial. The treatment phase will consist of 44 treatments over thirteen weeks. The acute treatment phase will consist five daily treatments over the course of six weeks, followed by twice weekly continuation treatments for seven weeks. Responders will be eligible to enter the durability phase. For assessment of durability, responders will be assessed quarterly for up to one year from the end of the treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Males and females, 18-88 years of age
* Diagnosed as suffering from OCD according to the DSM-V.
* Subjects with a YBOCS score of >20.
* If on SRI, patient must be maintained on current dosages (with or without additional antidepressant or psychotropic augmentation for treatment of OCD), at a stable therapeutic dosage for at least 2 months prior to study entry and for the duration of the trial.
* If in CBT, must be in the maintenance stage (i.e., not receiving active training in exposure and response prevention, which is the core component of this treatment). CBT can be with teletherapy but must be for a minimum of ten sessions with a symptom checklist, hierarchy, with exposure and response prevention therapy.
* Have negative or justified responses by the investigator to all questions listed on the Transcranial Magnetic Stimulation Safety Screening questionnaire (TASS).
* According to the treating physician the subject is compliant with taking medication, if applicable.
* Subject is capable and willing to provide informed consent and assent.
* Willing and able to adhere to the treatment schedule.
* Must own a smartphone.
* All comorbid diagnoses have been stable for 3 months and anticipated to be stable for the 3 months treatment duration.

Exclusion Criteria:

* Subjects diagnosed as suffering from any other Axis I diagnosis as the primary diagnosis.
* Comorbid, secondary psychiatric diagnoses are unstable and are likely to require changes in therapeutic regimens even if OCD improves.
* Present suicidal risk as assessed by the investigator using the Columbia Suicide Severity Rating Scale, brief mental status exam and psychiatric interview or a history of attempted suicide in the past year.
* History of epilepsy or seizure (EXCEPT those therapeutically induced by ECT and febrile seizures in infancy).
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure, or history of significant head trauma with loss of consciousness for greater than or equal to 5 minutes.
* History of head injury necessitating cranial surgery or prolonged coma.
* History of any ferromagnetic of conductive material in the head including the eyes and ears (outside the mouth).
* Known history of any metallic particles in the eye, implanted neurostimulators, intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes).
* History of significant hearing loss.
* Subjects with significant neurological disorder or insult including, but not limited to
* Any condition likely to be associated with increased intracranial pressure
* Space occupying brain lesion
* History of cerebrovascular accident
* Transient ischemic attack within two years
* Cerebral aneurysm
* Multiple sclerosis
* Substance use disorder within the past 6 months (except nicotine and caffeine).
* Currently participating in another therapeutic clinical study.
* Suffer from an unstable physical, systemic and metabolic disorder such as unstable blood pressure, unstable blood sugar, or acute, unstable cardiac disease.
* Subject on high doses of antidepressant or psychotropic medications, which are known to lower the seizure threshold. Subject is currently on Clomipramine.
* Significant possibility of death within eighteen months of baseline.
* Planned surgeries that will interrupt the study schedule within eighteen months of baseline
* Treatment with any TMS in the past year.
* Women who are breast-feeding.
* Women who are pregnant or with suspected pregnancy.
* Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale (YBOCS) | 6 weeks
  Change in YBOCS scores from baseline to the end of six weeks between the active Deep TMS and Sham treatment groups.
  Scores on the YBOCS range from 0 (no Symptoms) to 40 (Extreme Symptoms).
Yale Brown Obsessive Compulsive Scale (YBOCS) | 13 weeks
  Change in YBOCS scores from baseline to the end of thirteen weeks between the active Deep TMS and Sham treatment groups.
  Scores on the YBOCS range from 0 (no Symptoms) to 40 (Extreme Symptoms).